CLINICAL TRIAL: NCT06587789
Title: A Multi-center, Prospective and Observational Study of Ribociclib in Combination With Adjuvant Endocrine Therapy for Patients With Early High-risk HR+HER2- Breast Cancer
Brief Title: Ribociclib in Combination With Adjuvant Endocrine Therapy for Patients With Early High-risk HR+HER2- Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The First Affiliated Hospital of Bengbu Medical University (Other); Jinhua Central Hospital (Other); Taizhou Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); The Affiliated People's Hospital of Ningbo University (Other Government); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); First People's Hospital of Hangzhou (Other); Affiliated Zhoushan Hospital of Wenzhou Medical University (Other); Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0726
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: Ribociclib; Breast Cancer; Adjuvant Endocrine Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ribociclib combined with endocrine therapy group: Patients with early high-risk HR+HER2- breast cancer will receive ribociclib (at a dose of 400mg per day for 3 weeks, followed by 1 week off, 4 weeks for 1 cycle) plus physician-selected endocrine therapy as adjuvant therapy. During three years of follow-up, their relevant clinical data will be recorded.
  Interventions: Drug: Ribociclib

INTERVENTIONS:
Drug: Ribociclib — Participants will receive ribociclib (at a dose of 400mg per day for 3 weeks, followed by 1 week off, 4 weeks for 1 cycle) plus physician-selected endocrine therapy (according to standard clinical practice, TAM or AI, with or without OFS).

SUMMARY:
The goal of this observational study is to learn about the effects of using ribociclib in combination with physician-selected endocrine therapy as adjuvant therapy for patients with early high-risk HR+HER2- breast cancer. The main question it aims to answer is:

Whether it is effective and safe to use ribociclib in combination with physician-selected endocrine therapy as adjuvant therapy for patients with early high-risk HR+HER2- breast cancer? Participants will receive ribociclib (at a dose of 400mg per day for 3 weeks, followed by 1 week off, 4 weeks for 1 cycle) plus physician-selected endocrine therapy for three years. During the follow-up, their relevant clinical data will be recorded.

DETAILED DESCRIPTION:
In this multi-center, prospective and observational study, we aim to learn about the efficacy and safety of using ribociclib in combination with physician-selected endocrine therapy as adjuvant therapy for patients with early high-risk HR+HER2- breast cancer. After being evaluated by the researchers as early high-risk HR+HER2- breast cancer patients, signing the informed consent, and being screened to meet the inclusion criteria, eligible participants will be enrolled to receive ribociclib (at a dose of 400mg per day for 3 weeks, followed by 1 week off, 4 weeks for 1 cycle) plus physician-selected endocrine therapy. During there years of follow-up, their relevant clinical data will be recorded.

Enrolled patients are recommended to receive 3 years of ribociclib combined with ET, or until evidence of disease recurrence is observed or other discontinuation criteria are met (whichever occurs earliest).

ET will be administered during the observational phase of the study (3 years) according to the prescription selected by the physician. At the end of the research observation phase, according to medical indication, standard adjuvant ET should continue for 2-8 years, and the total treatment duration can be up to 10 years.

According to physician's choice, participants use the approved standard adjuvant ET (e.g., according to standard clinical practice, TAM or AI, with or without OFS). Fulvestrant should not be used for adjuvant therapy at any time during the study period.

Review of imaging (ultrasound,CT or MRI) of common recurrent sites throughout the body every 3 months before and after dosing, and every 6 months after 2 years until disease recurrence or death or the end of this study. This is the current follow-up interval recommended by the Chinese Anticancer Association Breast Cancer Diagnosis and Treatment Guidelines and Specifications, Version 2024, which does not increase the burden of follow-up for patients.

Records of blood-related indicators (according to the instructions of ribociclib) (blood routine, biochemical indicators) were reviewed during the treatment follow-up. Medical staff, graduate students, and technicians complete the record of the patient-reported outcomes (PROs) (pre-drug and 1,3,6,12,18,24,36 months post-drug) in real time through mutiple questionnaire survey such as WeChat applets, phone calls, text messaging, and face-to-face visits.

The study will collect primary and recurrent metastatic tumor tissues and blood, using multi-gene detection, proteomic and other means to detect samples, and explore the biomarkers associated with ribociclib treatment.

This study is expected to have an enrollment time of 24 months and a follow-up time of 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Before any trial-related procedures, sign a written informed consent, and be willing and able to follow the planned visits, research treatment, laboratory examination and other test procedures;
2. Age 18-80 years old, female (both pre/post menopausal);
3. The patient's initial diagnostic tissue specimens were confirmed to be HR+, HER2- early high-risk invasive breast cancer without evidence of disease recurrence or distant metastasis.
4. The patient must have undergone radical surgery for the primary breast tumor. The cut edge of the removed specimen must be free from histological tumor residue (including invasive breast cancer or ductal carcinoma in situ [DCIS]). If supraclavicular or internal breast lymph nodes are considered for metastasis but cannot be surgically removed, radiotherapy should be carried out in the remaining lymph node drainage area in accordance with local guidelines.
5. After surgical resection, the tumor was completely removed, and there was no tumor at the end of the surgical specimen microscope, and it belonged to one of the following stages:

   * Pathological Stage IIB or III
   * Pathological Stage IIA as listed below:
   * N1 or N0, and: grade 3, or grade 2, meeting any of the following criteria:

   ( Ki67 ≥ 20%, or Oncotype DX breast recurrence score ≥ 26, or MammaPrint classification of high risk)

   Attention:
   * For patients with tumor anatomical stage IIA N0: Patients are ineligible if Grade 1 or Unknown (Gx).
   * Patients receiving neoadjuvant therapy must meet the above criteria in any preoperative staging/samples and/or surgical specimens (for staging, if Stage IIA, N0, also including grading and Ki67 or gene expression testing).
   * AJCC 8th edition anatomic staging requirements determine T, N, and M categories. ALND is the preferred method for axillary lymph node staging; however, SLN dissection may be used to determine N classification in the following situations: No metastasis in the SLN (patients are considered as pN0); Slight metastasis in the SLN (patient considered as pN1mi); Patients with T1-2 and no clinically significant nodes before surgery, no neoadjuvant chemotherapy, at least 1 macrometastasis in 1 or 2 SLNs, no clustered swollen lymph nodes or severe extra-lymph node diseases during SLN clearance (patients are considered as pN1).
6. A maximum of 12 months from surgery to enrollment.
7. Patients with an ECOG score of ≤3, allowing the combination of other asymptomatic underlying diseases.
8. The patient can swallow oral endocrine drugs, regardless of the type of endocrine drugs.
9. The patient agrees to take paraffin samples from the primary lesions (including the primary lesions and lymph nodes), tumor tissue and blood samples from the recurrent lesions for future exploratory biomarker analyses
10. The patient has completed (neo)adjuvant chemotherapy and standard radiotherapy (when indicated) in accordance with clinical practice guidelines.

Exclusion Criteria:

1. The patient has received any CDK4/6 inhibitors in the past.
2. Metastatic diseases (including contralateral axillary lymph nodes)
3. Patients have received ET (tamoxifen or aromatase inhibitors or raloxifene) for the prevention of breast cancer.
4. Unwilling to participate in the quality of life questionnaire score or provide tissue samples at the time of recurrence

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population who meet the above mentioned inclusions will be selected from cooperative hospitals.
Sampling Method: Probability Sample
Enrollment: 286 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival(iDFS) | 3 years
  iDFS using STEEP criteria (Standardized Definitions for Efficacy End Points in Adjuvant Breast Cancer Trials), as assessed by Investigator. iDFS is defined as time from the date of randomization to the date of the first event of local invasive breast recurrence, regional invasive recurrence, distant recurrence, death (any cause), contralateral invasive BC, or second primary non-breast invasive cancer (excluding basal and squamous cell carcinomas of the skin).

SECONDARY OUTCOMES:
Distant recurrence-free survival(DRFS) | 3 years
  DRFS is defined as the time from date of randomization to date of first event of distant recurrence, or death (any cause).
Distant disease-free survival(DDFS) | 3 years
  DDFS using STEEP criteria. DDFS is defined as the time from date of randomization to date of first event of distant recurrence, death (any cause), or second primary non-breast invasive cancer (excluding basal and squamous cell carcinomas of the skin).
Overall Survival | 3 years
  OS is defined as the time from date of randomization to date of death due to any cause.
Frequency of AE/SAE | 3 years
  Adverse Events assessed by investigator (type, frequency, severity (graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.5.0)), seriousness)
Quality of life by the Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline and 1,3,6,12,18,24,36 months after therapy
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The EORTC QLQ-C30 contains functional scales, symptom scales, single items scale and a global health status/QoL scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life by the Quality of Life Questionnaire - Breast cancer module (QLQ-BR23) | At baseline and 1,3,6,12,18,24,36 months after therapy
  This EORTC breast cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BR23 contains 23 items incorporating five multi-item scales to assess systemic therapy side effects, arm symptoms, breast symptoms, body image and sexual functioning. All of the scales and single-item measures range in score from 0 to 100. Higher scores typically indicate better quality of life, while lower scores may suggest poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China